CLINICAL TRIAL: NCT03746925
Title: Randomized Control Trial Comparing Short-term Outcomes After Direct Anterior and SuperPATH Approaches
Brief Title: Comparing Short-term Outcomes After Direct Anterior and SuperPATH Hip Arthroplasty Approaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SuperPATH
Record Dates: First submitted 2018-11-09; First posted 2018-11-20 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: DAA; SuperPATH; Direct Anterior Approach; THA

STUDY DESIGN:
Intervention Model Description: It is a 2 group, parallel study where they will be randomized into one of the two groups. One will receive SuperPATH approach and the other will receive DAA.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Anterior Approach (DAA) (Active Comparator): Direct Anterior Approach surgery to replace the hip.
  Interventions: Procedure: Direct Anterior Approach (DAA)
- SuperPATH (Experimental): SuperPATH approach surgery to replace the hip.
  Interventions: Procedure: SuperPATH

INTERVENTIONS:
Procedure: Direct Anterior Approach (DAA) — Direct Anterior Approach surgery to replace the hip.
  Arms: Direct Anterior Approach (DAA)
Procedure: SuperPATH — SuperPATH approach surgery to replace the hip.
  Arms: SuperPATH

SUMMARY:
This study involves comparing the outcomes after using the Direct Anterior Approach (DAA) and the Supercapsular Percutaneously Assisted Total Hip (SuperPATH) approach. These are two approaches to hip replacement that both replace hips without cutting any muscles. DAA approach has been used for many years, but it has a high learning curve and can be difficult for doctors to use, it is however linked with fewer complications when performed by an experienced doctor. SuperPATH is a newer technique which has been shown in studies to be adopted with less complications even during the learning phase. It also shows cost-saving results, showing a reduced length of stay for patients and better 30-day readmission rates. There is pressure on surgeons, from both patients and administration to use techniques that spare tissue, offer early functionality without compromising long-term outcomes. The SuperPATH can meet this benchmark but uptake has been slow, the investigators believe that it is due to the learning curve shown by this approach. The senior surgeon at The Ottawa Hospital is experienced in both techniques, using a trial the investigators can compare the two techniques and help encourage surgeons to change to a procedure that has demonstrated a low complication profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral THA
* Over 18 years of age and below 80
* Subject is willing and able to complete required study visits and assessments
* Subject is willing to sign the approved informed consent form

Exclusion Criteria:

* Subject has both a body mass index (BMI) and waist circumference measurements greater than 35.0kg/m2 and 102.0cm, respectively for men, and 35.0kg/m2 and 88.0cm, respectively for women at screening
* Subject is currently enrolled in another clinical investigation related to lower limbs, which could affect the endpoints of this protocol
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
* Subject is currently incarcerated or has impending incarceration
* Previous hip surgery or infection on ipsilateral hip

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-07 (Actual); Primary Completion 2023-01-07 (Estimated); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hip disability and Osteoarthritis Outcome Score (HOOS) activities of daily living (ADL) | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  This asks the patient how their hip functions during their daily life. It has 5 subscales measuring Pain, Symptoms, ADL, Sports/Recreation and Quality of Life (which is calculated using all the subscores). Each subscale is calculated using the mean score, with each score range being from 0 to 4. The subscore is normalized such that the lower the number the more extreme the problem is. To calculate Quality of Life, the mean of the other 4 subscores are taken to calculate the score.
Change in Gait analysis | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  This is done by a biomechanics lab for a subsection of 30 patients to test their hip movements.

SECONDARY OUTCOMES:
Change in EQ-5D-5L | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  Generic health status. Each question is scored from 1-5, with 1 being no problems and 5 being severe problems. These scores are not aggregated. There are 5 questions, mobility, self-care, usual activities, pain and anxiety. The last page is asking the participant to self score their health that day out of 100.
Change in Pre-post Hgb | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 2 weeks post-operatively.
  Checks blood oxygen level
Change in Visual Analog Scale (VAS) Pain Score | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 2 weeks post-operatively.
  To measure pain. This is a line with left most end representing no pain with the rightmost representing extreme pain. The participant puts a line where they feel that day and it is measured with a ruler to determine score out of 100. The line is 100mm long.
Change in Complication rates | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  Complications such as fractures that the participant experiences will be assessed
Readmission rates | 3 months post-operatively
  Any readmission rates for the participant
Change in Timed-up-and-go (TUG) | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  The time it takes for the participant to get up from a chair walk 3 metres forward and back and sit back down
Change in Timed-Stair-Climb (TSC) | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  The time it takes for a participant to go up and down a flight of 10 stairs.
Change in Range of Motion (ROM) | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  IR and ER ROM at flexion and extension, this is measured using a goniometer (which is an instrument that measures an angle).
Change in X-rays (AP pelvis & lateral) | This is from baseline (can be measured anytime to a maximum of one month before surgery) to 12 months post-operatively.
  To check how their bones are faring in their hip area

CONTACTS AND LOCATIONS:
Overall Officials: Wade Gofton, MD, FRCSC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
To keep patient confidentiality safe.

REFERENCES:
- [Background] Chow J, Penenberg B, Murphy S. Modified micro-superior percutaneously-assisted total hip: early experiences & case reports. Curr Rev Musculoskelet Med. 2011 Sep;4(3):146-50. doi: 10.1007/s12178-011-9090-y. PMID 21789576
- [Background] Della Torre PK, Fitch DA, Chow JC. Supercapsular percutaneously-assisted total hip arthroplasty: radiographic outcomes and surgical technique. Ann Transl Med. 2015 Aug;3(13):180. doi: 10.3978/j.issn.2305-5839.2015.08.04. PMID 26366397
- [Background] Gofton W, Chow J, Olsen KD, Fitch DA. Thirty-day readmission rate and discharge status following total hip arthroplasty using the supercapsular percutaneously-assisted total hip surgical technique. Int Orthop. 2015 May;39(5):847-51. doi: 10.1007/s00264-014-2587-4. Epub 2014 Nov 16. PMID 25398472
- [Background] Chow J, Fitch DA. In-hospital costs for total hip replacement performed using the supercapsular percutaneously-assisted total hip replacement surgical technique. Int Orthop. 2017 Jun;41(6):1119-1123. doi: 10.1007/s00264-016-3327-8. Epub 2016 Nov 12. PMID 27838761
- [Background] SMITH-PETERSEN MN, LARSON CB, et al. Complications of old fractures of the neck of the femur; results of treatment of vitallium-mold arthroplasty. J Bone Joint Surg Am. 1947 Jan;29(1):41-8. No abstract available. PMID 20284684
- [Background] Judet J, Judet H. [Anterior approach in total hip arthroplasty]. Presse Med. 1985 May 4;14(18):1031-3. French. PMID 3158949
- [Background] Kennon RE, Keggi JM, Wetmore RS, Zatorski LE, Huo MH, Keggi KJ. Total hip arthroplasty through a minimally invasive anterior surgical approach. J Bone Joint Surg Am. 2003;85-A Suppl 4:39-48. doi: 10.2106/00004623-200300004-00005. No abstract available. PMID 14652392
- [Background] Bal BS, Vallurupalli S. Minimally invasive total hip arthroplasty with the anterior approach. Indian J Orthop. 2008 Jul;42(3):301-8. doi: 10.4103/0019-5413.41853. PMID 19753156
- [Background] Barrett WP, Turner SE, Leopold JP. Prospective randomized study of direct anterior vs postero-lateral approach for total hip arthroplasty. J Arthroplasty. 2013 Oct;28(9):1634-8. doi: 10.1016/j.arth.2013.01.034. Epub 2013 Mar 19. PMID 23523485
- [Background] Goebel S, Steinert AF, Schillinger J, Eulert J, Broscheit J, Rudert M, Noth U. Reduced postoperative pain in total hip arthroplasty after minimal-invasive anterior approach. Int Orthop. 2012 Mar;36(3):491-8. doi: 10.1007/s00264-011-1280-0. Epub 2011 May 25. PMID 21611823
- [Background] Alecci V, Valente M, Crucil M, Minerva M, Pellegrino CM, Sabbadini DD. Comparison of primary total hip replacements performed with a direct anterior approach versus the standard lateral approach: perioperative findings. J Orthop Traumatol. 2011 Sep;12(3):123-9. doi: 10.1007/s10195-011-0144-0. Epub 2011 Jul 12. PMID 21748384
- [Background] Nakata K, Nishikawa M, Yamamoto K, Hirota S, Yoshikawa H. A clinical comparative study of the direct anterior with mini-posterior approach: two consecutive series. J Arthroplasty. 2009 Aug;24(5):698-704. doi: 10.1016/j.arth.2008.04.012. Epub 2008 Jun 13. PMID 18555653
- [Background] Anterior Total Hip Arthroplasty Collaborative Investigators; Bhandari M, Matta JM, Dodgin D, Clark C, Kregor P, Bradley G, Little L. Outcomes following the single-incision anterior approach to total hip arthroplasty: a multicenter observational study. Orthop Clin North Am. 2009 Jul;40(3):329-42. doi: 10.1016/j.ocl.2009.03.001. PMID 19576400
- [Background] Xie J, Zhang H, Wang L, Yao X, Pan Z, Jiang Q. Comparison of supercapsular percutaneously assisted approach total hip versus conventional posterior approach for total hip arthroplasty: a prospective, randomized controlled trial. J Orthop Surg Res. 2017 Sep 25;12(1):138. doi: 10.1186/s13018-017-0636-6. PMID 28946892
- [Background] Meermans G, Konan S, Das R, Volpin A, Haddad FS. The direct anterior approach in total hip arthroplasty: a systematic review of the literature. Bone Joint J. 2017 Jun;99-B(6):732-740. doi: 10.1302/0301-620X.99B6.38053. PMID 28566391
- [Background] Lachin JM, Matts JP, Wei LJ. Randomization in clinical trials: conclusions and recommendations. Control Clin Trials. 1988 Dec;9(4):365-74. doi: 10.1016/0197-2456(88)90049-9. PMID 3203526
- [Background] Ehrich EW, Davies GM, Watson DJ, Bolognese JA, Seidenberg BC, Bellamy N. Minimal perceptible clinical improvement with the Western Ontario and McMaster Universities osteoarthritis index questionnaire and global assessments in patients with osteoarthritis. J Rheumatol. 2000 Nov;27(11):2635-41. PMID 11093446
- [Background] Gofton W, Fitch DA. In-hospital cost comparison between the standard lateral and supercapsular percutaneously-assisted total hip surgical techniques for total hip replacement. Int Orthop. 2016 Mar;40(3):481-5. doi: 10.1007/s00264-015-2878-4. Epub 2015 Jul 9. PMID 26156723
- [Background] Varin D, Lamontagne M, Beaule PE. Does the anterior approach for THA provide closer-to-normal lower-limb motion? J Arthroplasty. 2013 Sep;28(8):1401-7. doi: 10.1016/j.arth.2012.11.018. Epub 2013 Mar 16. PMID 23507070
- [Background] Kerrigan DC, Todd MK, Della Croce U. Gender differences in joint biomechanics during walking: normative study in young adults. Am J Phys Med Rehabil. 1998 Jan-Feb;77(1):2-7. doi: 10.1097/00002060-199801000-00002. PMID 9482373
- [Background] Judge JO, Ounpuu S, Davis RB 3rd. Effects of age on the biomechanics and physiology of gait. Clin Geriatr Med. 1996 Nov;12(4):659-78. PMID 8890109